CLINICAL TRIAL: NCT04027881
Title: Improving Print Knowledge for Children With Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: tambyraja.1
Record Dates: First submitted 2019-06-28; First posted 2019-07-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to start the intervention immediately after baseline assessment (i.e., treatment) or approximately 15 weeks later after the baseline assessment (i.e., waitlist control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAR - immediate (Experimental): Receive 15-week STAR intervention immediately after pretest.
  Interventions: Behavioral: Sit Together and REad
- STAR - waitlist control (No Intervention): No intervention for the 15 weeks after pretest.

INTERVENTIONS:
Behavioral: Sit Together and REad — STAR is an evidence-based home-based shared book reading intervention designed to improve the foundational reading skills of preschoolers who are at risk for reading disabilities.
  Other Names: STAR
  Arms: STAR - immediate

SUMMARY:
This R56 award will address questions pertaining to the feasibility of the Sit Together and Read (STAR) intervention for children with hearing loss (HL). Evidence suggests that STAR, a caregiver-implemented early literacy intervention, imparts positive effects on print knowledge gains and later reading outcomes for children at risk for reading difficulties, such as those with language impairment and those living in poverty. To date there are no large-scale studies examining literacy interventions for children with HL, who are also known to be at risk for reading disorders. However, prior to engaging in a large-scale study, this research will establish preliminary feasibility and efficacy data for this specific population who will likely benefit from a evidence-based, manualized intervention. In addition to collecting pilot data regarding the feasibility and efficacy of this intervention for children with HL, this study will also determine barriers and challenges experienced by caregivers of children with HL in implementing the intervention. As such, this study will also yield important information regarding adaptations of the existing STAR intervention that may be required for successful and effective implementation for children with HL, and can be incorporated into future submissions.

DETAILED DESCRIPTION:
This study will use a randomized (1:1) waitlist controlled trial design to test the effects of a 15-week caregiver-implemented STAR intervention for children with HL. STAR incorporates a high intensity of home-based shared book reading sessions (i.e., 4 times a week) in which caregivers embed guided discussions about foundational reading concepts that are prerequisites for learning to read. Caregivers will receive individualized training and materials for implementing STAR at home with their child. Caregivers will be provided with materials and equipment to read and audio record their readings 4 times a week, and to engage in meaningful, instructional dialogue while reading, in order to help children learn about foundational reading topics, such as letter names and sounds.

The study is guided by the following specific aims: Aim 1: Determine the extent to which caregivers of children with HL can effectively implement a home-based reading intervention for their children. Hypothesis 1: Caregivers will effectively implement the STAR intervention but there will be some variability. Aim 2: Improve the early literacy skills of children with HL, by implementing STAR. Hypothesis 2: Children whose caregivers are randomized to the home-implemented STAR intervention will demonstrate significantly greater gains in early reading skills over the implementation period, compared to those randomized to a waitlist control condition. Aim 3: Identify implementation barriers or challenges experienced by caregivers of children with HL. This aim is exploratory and will inform potential adaptations to the intervention that may be required for future, more successful intervention implementation by caregivers of children with HL.

Upon completion, the investigators will have established the feasibility and effectiveness of the STAR intervention for children with HL and their caregivers. Data from this study will be the foundation for a large-scale randomized-controlled clinical trial that focuses on improving the reading outcomes of children with a range of communication disorders and identifying optimal methods for supporting their caregivers.

ELIGIBILITY:
Inclusion Criteria for children:

* Child 4 years, 0 months to 5 years, 11 months at enrollment
* Child has bilateral sensorineural hearing loss
* child has at least one years' experience of hearing device use (hearing aid, cochlear implant)
* child does not have a severe cognitive disability

Inclusion Criteria for caregivers:

* Caregiver willing to attend in-person meetings
* Caregiver willing to read regularly to the child in English for 15 consecutive weeks

Exclusion Criteria:

-

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
STAR Log | 15-week intervention period
  Document intensity, defined as occurrence and length of each session and targeted goals within each.
STAR Fidelity Coding Checklist (FCC) | 15-week intervention period
  Document dosage, defined as the volume of explicit targeting of print-related objectives during STAR sessions.
Preschool Word and Print Awareness (PWPA) | 15-week intervention period
  Examines knowledge of 15 print concepts. Scores on this scale range from 0-17, with higher scores indicative of better performance.
Phonological Awareness Literacy Screening-PreK (PALS-PreK) | 15-week intervention period
  Upper and Lower Case Letter Knowledge subtests will identify the number of letters children can name. The range on these subtests is 0-26, with higher scores indicative of better performance. The name writing subtest will assess children's ability to write their own name. The range on this subtest is 0-7, with higher scores indicative of better performance.
Test of Preschool Emergent Literacy (TOPEL) | 15-week intervention period
  The print knowledge subtest will be used to assess children's skills on a variety of print-related tasks, such as distinguishing print from other visual stimuli and identifying alphabet letters. Raw scores on this subtest range from 0-36, with higher scores indicative of better performance

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No